CLINICAL TRIAL: NCT05796830
Title: Determination of the Effect of Puzzle Use on Cognitive Functions, Surgical Recovery and Quality of Life in Elderly Patients Undergoing Orthopedic Surgery
Brief Title: Determination of the Effect of Puzzle Use in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, Assoc. Prof, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22-106
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Quality of Life; Surgery; Postoperative Confusion; Cognitive Dysfunction
Keywords: Postoperative Recovery, Cognitive Function, Surgery, Quality of Life, Elderly Patient
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This studyis a single-center and randomized controlled clinical trial. Patients who accepted to participate in the study and met the inclusion criteria will be assigned to the intervention (n= 35) or control group (n= 35) according to the computer- based randomization table.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Before the operation, the rules of the puzzle will be explained to the patients in the intervention group and how it will be applied will be shown. Then, Patient Diagnosis Form, Mini-Mental State Test and Quality of Life Scale will be administered.On the 1st, 2nd and 3rd days after the surgery, the rules of the puzzle will be reminded again and the puzzle will be applied to the patients once a day. After the puzzle application on the 1st, 2nd and 3rd days after the surgery, the Mini-Mental State Test will be applied to the patients. Postoperative Recovery Index and Quality of Life Scale will be applied on the 3rd postoperative day.
  Interventions: Other: Puzzle application
- Control Group (No Intervention): Patients in the control group will be followed according to routine clinical procedure. Since there are no procedures or interventions in clinical procedures, only patient monitoring will be performed. The patients in the control group will also be followed and evaluated with the same forms at the same time.

INTERVENTIONS:
Other: Puzzle application — Five expert opinions will be taken for the puzzle application to be applied after the surgery, and the application and difficulty level of the puzzle will be decided.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to determine the effects of the use of a simple, reliable and cost-effective puzzle on post-operative cognitive function changes, postoperative recovery, and quality of life using questionnaires and face-to-face interview techniques.

DETAILED DESCRIPTION:
Aging is a process involving biological, physiological and psychological changes. With aging, deterioration in brain, behavior and cognitive functions is observed. In this process, physical and cognitive deficiencies and slow thinking can be seen. The independence of elderly individuals in meeting their self-care decreases. Over time, individuals become unable to meet their needs and this reduces the quality of life of individuals. With the developing technology, perioperative care techniques began to develop and the number of surgical procedures applied to elderly patients began to increase.One of the most important goals in the field of health today and in the future will be to increase the quality of life of individuals. It is becoming increasingly important to determine the effective factors to protect cognitive functions in elderly individuals.After surgical procedures, patients may experience memory loss and decrease in concentration. Symptoms indicating a decrease in cognitive functions were named as postoperative cognitive dysfunction. Compared to other individuals undergoing surgery, the rate of cognitive changes in the early period is higher in the elderly.Especially, elderly patients who underwent orthopedic surgery are thought to be a risky patient group for postoperative cognitive impairment.Solving jigsaw puzzles is a low-cost, motivating, visuospatial cognitive-challenging activity.This study will be conducted in order to determine the effect of this strain on the cognitive functions of the individual and to investigate the effect of focusing on completing the puzzle on post-operative recovery and quality of life, as it will focus the individual's perception on a certain point.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older,
* Having been hospitalized in the orthopedic service for at least three days after the operation,
* Having undergone orthopedic surgery,
* No hearing or vision problems,
* Able to communicate,
* No cognitive or psychiatric problems,
* At least primary school graduate,
* Patients who agreed to participate in the study

Exclusion Criteria:

* Using jigsaw puzzles regularly,
* Using drugs that affect memory and thinking

These drugs are:

1. Sedative and Hypnotic Drugs

   * Benzodiazepines
   * Barbiturates
   * Non-barbiturate
   * Other Sedative and Hypnotics (zolpidem, buspirone, hydroxyzine)
2. Anticonvulsant Drugs
3. Drugs Used in Parkinson's Treatment
4. Drugs Used in the Treatment of Psychiatric Diseases
5. Drugs with Narcotic Analgesic Effects
6. Anesthetic Drugs
7. Neuromuscular Blocking Drugs - Patients with cerebrovascular accident or head injury

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-28 (Estimated); Primary Completion 2023-10-29 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Change of Cognitive Function by the Standardized Mini-Mental Test | 1st, 2nd and 3rd days after the surgery
  1st, 2nd and 3rd days after the surgery, the puzzle will be applied to the patients once a day. Then the Standardized Mini-Mental Test will be applied to the patients.This test is a measurement tool that can be easily administered within 5-10 minutes, does not include questions about mental processes, and focuses only on cognitive processes.The Standardized Mini Mental Test consists of 11 items under 5 main headings: orientation (10 points), attention and calculation (5 points), recording (3 points) and recall memory (3 points) and language (9 points). It is evaluated out of 30 points. The increase in the score obtained from the test indicates that the severity of cognitive destruction decreases.
Change of Postoperative Recovery by the Postoperative Recovery Index | 3rd day after the surgery
  Postoperative Recovery Index will be applied on the 3rd postoperative day. Postoperative Recovery Index consists of 5 sub-dimensions and 25 items. Sub dimensions; psychological symptoms, physical activities, general symptoms, intestinal symptoms, and craving-desire symptoms. While determining the sub-dimension score, the scores of the related items are summed and their arithmetic averages are taken. For the total score; All items are summed and the arithmetic average is taken. It states that the higher the scores obtained from the index, the more difficulty in post-operative recovery, and the easier the post-operative recovery as the scores decrease.
Change of Quality of Life by Quality of Life Scale in Older People (CASP-19) | 3rd day after the surgery
  Quality of Life Scale in Older People (CASP-19) will be applied on the 3rd postoperative day. The scale consists of 19 items and four sub-dimensions. These sub-dimensions are control, autonomy, pleasure, and self-actualization. Each item of the original scale was graded as a 4-point Likert-type scale ranging from "never" (0 points) to "always" (3 points). Scale items are scored between 0 and 3 points. An increase in the score obtained from the scale indicates an increase in the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Emel Çanakçı, RN, Principal Investigator — Saglik Bilimleri Universitesi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rundshagen I. Postoperative cognitive dysfunction. Dtsch Arztebl Int. 2014 Feb 21;111(8):119-25. doi: 10.3238/arztebl.2014.0119. PMID 24622758
- [Background] Fissler P, Kuster OC, Loy LS, Laptinskaya D, Rosenfelder MJ, von Arnim CAF, Kolassa IT. Jigsaw Puzzles As Cognitive Enrichment (PACE) - the effect of solving jigsaw puzzles on global visuospatial cognition in adults 50 years of age and older: study protocol for a randomized controlled trial. Trials. 2017 Sep 6;18(1):415. doi: 10.1186/s13063-017-2151-9. PMID 28877756